CLINICAL TRIAL: NCT04199234
Title: A Randomized, Double Blind, Crossover Study to Compare the Tolerability of Microencapsulated Iron Compared to a Conventional Iron Supplement in the Market
Brief Title: A Study to Compare the Tolerability of Microencapsulated Iron Compared to a Conventional Iron Supplement in the Market
Acronym: IRON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: UCAMCFE-0011
Record Dates: First submitted 2019-12-10; First posted 2019-12-13 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2020-03

CONDITIONS: Supplement
MeSH Terms: interventions — Iron-Dextran Complex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): 60 mg Encapsulated Iron
  Interventions: Dietary Supplement: Experimental product consumption
- control group (Active Comparator): 60 mg Iron sulphate
  Interventions: Dietary Supplement: Comparator product consumption (Iron sulphate)

INTERVENTIONS:
Dietary Supplement: Experimental product consumption — Consumption of an encapsulated iron supplement, 60 mg iron per day over 14 days, 2 hours before lunch
  Arms: experimental group
Dietary Supplement: Comparator product consumption (Iron sulphate) — Consumption of iron supplement, 60 mg iron per day over 14 days, 2 hours before lunch
  Arms: control group

SUMMARY:
The purpose of this study is to compare the frequency of appearance of the total clinical manifestations (expected adverse event: nausea, vomiting, heartburn, abdominal pain, gas/swelling, diarrhea, headache, shortness of breath, metallic taste and constipation) after consuming microencapsulated iron and comparator for 14 days.

DETAILED DESCRIPTION:
Subjects will consume a daily dose once per day for 14 days with a washout period of two menstrual cycles between the two products. After this washout period, subjects will return to the clinical and will undergo identical procedures with counter order of the intervention.

Each day of the study will be recorded in a diary by each subject. Participants will be requested not to change their regular life habits and diet during the entire study.

ELIGIBILITY:
Inclusion criteria:

* Healthy premenopausal women (Age: 18-50)
* Not anemic
* Normal Iron status: hemoglobin (>12 g/dL)
* Normal BMI (20-25 kg/m²)
* Normal blood profile at screening: Complete blood count, platelets, Glucose, HbA1c, Electrolytes (Na, K, Cl), AST, ALT, bilirubin, y-GT), Creatinine, eGFR, blood urea nitrogen, uric acid, Total protein (albumin/ globulin)
* Subject is in good physical health as established by medical history, vital signs, physical examination and electrocardiogram (ECG)
* Normal urine profile at screening: pH, protein, glucose, nitrite, ketone, bilirubin, urobilinogen, red blood cells, leukocytes, creatinine, sediments, absence of bacteria
* Regular menstrual cycle (28 +/- 5)
* Willingness not to change eating habits (do not start/ change of diet) and general habits (stop smoking) for the duration of the study
* C-reactive protein: < 5mg/L.

Exclusion Criteria:

* Previous participation in iron tolerability trials.
* Participation in a clinical research trial within 30 days prior to randomization
* Chronic medication (except oral contraceptives)
* Pregnancy or lactation
* Hb levels < 12g/dL (women) (anemia)
* Reported chronic disease
* Infectious disease
* Alcohol or drug abuse
* Hyperlipidemia as defined by LDL > 3.36 mmol/L (130 mg/dL) and/or triglycerides > 2.26 mmol/L (200 mg/dL).
* Relevant co-morbidities: Gastrointestinal disease such as peptic ulcer, enteritis, or ulcerative colitis, inflammation, pre-existing poorabsorption or liver disease, kidney disease, iron-storage disorders such as hemochromatosis, haemosiderosis, or chronic autoimmune inflammatory condition
* Serious illness that may confound study results or interfere with compliance
* Any other laboratory abnormality, medical condition or psychiatric disorder which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject
* Known intolerance to oral iron supplements
* Intake of iron suppl. and/or multivitamins containing iron during the last three months before study entry
* Use of any mineral/vitamin or other supplements during the past month prior to study
* Subject has a known allergy to the test material's active or inactive ingredients
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any active medical illness in last 48 h
* Sexually-active females who are not willing to use an effective form of birth control.
* Subjects with severe premenstrual symptoms (PMS)
* Subjects that have followed specific diet, eg. high protein diet, within 30 days prior to study start
* Previous gastric bypass, sleeve gastrectomy, or gastric band surgery
* Blood donation within the previous 1 months.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Frequency of appearance of the total clinical manifestations due to the consumption of both products | This variable will measure the changes in clinical manifestations during the period of each of the intakes, i.e., for 14 days, and during the washout period.
  The proportion of participants that reported at least one adverse event, which refers to the total of clinical manifestations due to the consumption of both products. Symptoms that were considered: nausea, heartburn, abdominal pain, gas/swelling, diarrhea, vomits, metallic taste, constipation, headache and respiratory distress.

SECONDARY OUTCOMES:
Frequency of appearance of each of the total clinical manifestations due to the consumption of both products | This variable will measure the changes in clinical manifestations during the period of each of the intakes, i.e., for 14 days, and during the washout period.
  The proportion of participants that reported at least one adverse event, which refers to each of the total of clinical manifestations due to the consumption of both products (individual symptoms that were considered: nausea, heartburn, abdominal pain, gas/swelling, diarrhea, vomits, metallic taste, constipation, headache and respiratory distress)
Change in the total number of incidences/complaints related to the study product | This variable will measure the changes in clinical manifestations during the period of each of the intakes, i.e., for 14 days, and during the washout period.
  Symptoms: nausea, heartburn, abdominal pain, gas/swelling, diarrhea, vomits, metallic taste, constipation, headache, and respiratory distress
Number of clinical manifestations that subjects experience | This variable will measure the changes in clinical manifestations during the period of each of the intakes, i.e., for 14 days, and during the washout period.
  Symptoms: nausea, heartburn, abdominal pain, gas/swelling, diarrhea, vomits, metallic taste, constipation, headache, and respiratory distress
Overall intensity of clinical manifestations that subjects experience (nausea, heartburn, abdominal pain, gas/swelling) | This variable will measure the changes in clinical manifestations during the period of each of the intakes, i.e., for 14 days, and during the washout period.
  Intensity was measured with VAS scale
Overall intensity of clinical manifestations that subjects experience (diarrhea and vomits) | This variable will measure the changes in clinical manifestations during the period of each of the intakes, i.e., for 14 days, and during the washout period.
  Intensity was measured with number of times.
Change in the acute intensity of adverse effects that subjects experience | This variable will measure the changes in clinical manifestations during the period of each of the intakes, i.e., for 14 days, and during the washout period.
  Symptoms: Nausea, heartburn, abdominal pain, gas/swelling, vomits, diarrhea, constipation, metallic taste, headache, and respiratory distress
Duration (number of days) of clinical manifestation | This variable will measure the changes in clinical manifestations during the period of each of the intakes, i.e., for 14 days, and during the washout period.
  This variable was measured in total duration (number of days) of symptom onset (symptoms: nausea, heartburn, abdominal pain, metallic taste, headache, diarrhea, constipation, gas/swelling, respiratory distress and vomits)
Duration (minutes per day) of clinical manifestation | This variable will measure the changes in clinical manifestations during the period of each of the intakes, i.e., for 14 days, and during the washout period.
  Daily duration (minutes) of symptom (nausea, heartburn, abdominal pain, gas, metallic taste, headache, and respiratory distress)
Health status using VAS scale | This variable will measure the changes in clinical manifestations during the period of each of the intakes, i.e., for 14 days, and during the washout period.
  Health status (daily and with respect to the previous day)
Physical activity | This variable will measure the changes in clinical manifestations during the period of each of the intakes, i.e., for 14 days, and during the washout period.
  Proportion of participants that experienced any impact on daily activity
Bowel movements | This variable will measure the changes in clinical manifestations during the period of each of the intakes, i.e., for 14 days, and during the washout period.
  Number of times subjects go to the toilet.
Stool morphology | This variable will measure the changes in clinical manifestations during the period of each of the intakes, i.e., for 14 days, and during the washout period.
  Stool type (Bristol scale)
Sleep quality | This variable will measure the changes in clinical manifestations during the period of each of the intakes, i.e., for 14 days, and during the washout period.
  Sleep quality measured on a scale of 1 to 5 (1 being poor sleep quality and 5 being very good sleep quality).
Sleep duration | This variable will measure the changes in clinical manifestations during the period of each of the intakes, i.e., for 14 days, and during the washout period.
  Number of hours subjects sleep
Ferritin | Day 1 and day 14 of each product consumption.
  Iron profile. By means of a blood draw.
Saturated transferrin | Day 1 and day 14 of each product consumption.
  Iron profile. By means of a blood draw.
Serum iron | Day 1 and day 14 of each product consumption.
  Iron profile. By means of a blood draw.
Hemoglobin | Day 1 and day 14 of each product consumption.
  Iron profile. By means of a blood draw.
Safety variables | Day 1 and day 14 of each product consumption.
  Safety parameters (physical examination, vital signs, blood and urine laboratory tests, adverse events other than expected in the study)

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No